CLINICAL TRIAL: NCT02189603
Title: Evaluation of Safety and Immunogenicity of Recombinant (E. Coli) Hepatitis E Vaccine（Hecolin®） in Seniors Aged Over 65 Years
Brief Title: Phase Ⅳ Clinical Trial of Recombinant Hepatitis E Vaccine（Hecolin®）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Xiamen Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor-Investigator, Jun Zhang, professor，Xiamen University, Xiamen University
Organization: Xiamen University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-HE-05
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis E
Keywords: hepatitis E; Immunogenicity; vaccine; safety
MeSH Terms: conditions — Hepatitis E | interventions — hecolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Senior group(over 65 years old)-HE (Experimental): Anti-HEV IgG seronegative participants over 65 years old were enrolled. Hepatitis E vaccine, containing 30mcg of HEV239 recombinant antigen adsorbed to alum adjuvant suspended in 0.5ml phosphate buffer, was given at 0, 1, 6m for three doses.
  Interventions: Biological: Recombinant (E. Coli) Hepatitis E Vaccine
- Younger groups(16-65 years old) (Active Comparator): Participants aged 16-65 years old were enrolled. Hepatitis E vaccine, containing 30mcg of HEV239 recombinant antigen adsorbed to alum adjuvant suspended in 0.5ml phosphate buffer, was given at 0, 1, 6m for three doses.
  Interventions: Biological: Recombinant (E. Coli) Hepatitis E Vaccine
- Senior group(over 65 years old)-Cont (No Intervention): Anti-HEV IgG seropositive participants over 65 years old were enrolled. This is the safety control group, without any intervention.

INTERVENTIONS:
Biological: Recombinant (E. Coli) Hepatitis E Vaccine
  Other Names: Hecolin®
  Arms: Senior group(over 65 years old)-HE; Younger groups(16-65 years old)

SUMMARY:
The purpose of this study is to determine the safety and immunogenicity of the recombinant hepatitis E vaccine in people older than 65 years, and evaluate the efficacy of hepatitis E vaccine in this population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people aged over 16 years old at the time of the first vaccination, normal intelligence and agree to sign the informed consent form.
* Healthy subjects as established by medical history and history-oriented clinical examination before entering into the study.
* Subjects will reside in the study region in the next 7 months.
* Free of history of hepatitis E.
* Can comply with the request of study.
* Axillary temperature is below 37 degree centigrade.

Exclusion Criteria:

For dose 1:

* receiving other vaccine or immunoglobulin within two weeks;
* Having serious allergic history to vaccine and medicine
* Eclampsia, epilepsy, encephalopathy and history of mental disease or family;
* Thrombocytopenia or other disturbance of blood coagulation which would lead to muscle injection taboo;
* Fixed or suspected deficiency of immunologic function, containing immunosuppressant treatment, genetic defect, HIV or other factors;
* Congenital malformation, eccyliosis or severe chronic disease;
* Fixed or suspected other disease including fever, active infection, liver and kidney disease, angiocardiopathy, malignancy, acute and chronic disease;
* joining other clinical study undergoing;
* women pregnant or in lactation.

For dose 2 or 3:

* Severe allergy for dose 1 or 2;
* Severe adverse reaction associated with last vaccination;
* New occurrence of symptoms meet dose 1 exclusion criteria after the first dose.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12-07 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-Serious Adverse Events | From month 0-7
  Any adverse events reported within one month post each vaccination would be recorded, any serious adverse events reported throughout the study would be recorded.

SECONDARY OUTCOMES:
anti-HEV IgG seropositive rate | at month 7
GMT of anti-HEV IgG | 7 month after first vaccination
  Serum sample would be collected at month 7, and geometric mean titer of anti-HEV IgG would be tested

CONTACTS AND LOCATIONS:
Locations (1):
- Center for disease control and prevention in Xiamen haicang district, Xiamen, Fujian, China

REFERENCES:
- [Background] Zhu FC, Zhang J, Zhang XF, Zhou C, Wang ZZ, Huang SJ, Wang H, Yang CL, Jiang HM, Cai JP, Wang YJ, Ai X, Hu YM, Tang Q, Yao X, Yan Q, Xian YL, Wu T, Li YM, Miao J, Ng MH, Shih JW, Xia NS. Efficacy and safety of a recombinant hepatitis E vaccine in healthy adults: a large-scale, randomised, double-blind placebo-controlled, phase 3 trial. Lancet. 2010 Sep 11;376(9744):895-902. doi: 10.1016/S0140-6736(10)61030-6. Epub 2010 Aug 20. PMID 20728932